CLINICAL TRIAL: NCT06607354
Title: The Effect of Consuming Grass Finished Lamb Meat on Omega-3 Blood Response Among Healthy Consumers
Brief Title: Consuming Grass Finished Lamb Improves Blood Plasma ω-3 Fatty Acid Response Among Healthy Consumers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Agri-Food and Biosciences Institute (Other)
Responsible Party: Principal Investigator, Lynda Perkins, Postdoctoral Researcher, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19.08v2
Record Dates: First submitted 2024-09-09; First posted 2024-09-23 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Lamb; Omega-3; Fatty acids; Plasma; Plasma phospholipids

STUDY DESIGN:
Intervention Model Description: Describe parallel arms
Who Masked: Participant
Masking Description: Describe it was the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentrate/ Cereal fed lamb (No Intervention): Participants to consume three portions of lamb per week for four consecutive weeks. The lamb diet was a concentrate/cereal pellet.
- Grass fed lamb (Experimental): Participants to consume three portions of lamb per week for four consecutive weeks. The lamb diet was grass only.
  Interventions: Other: Grass fed lamb

INTERVENTIONS:
Other: Grass fed lamb — This study investigated the impact of consuming grass finished lamb on total blood plasma and blood plasma phospholipids (PL) FA and on cardiovascular risk factors, including heart rate, blood pressure (BP), HDL-cholesterol, LDL-cholesterol, and TAG cholesterol, in humans.
  Arms: Grass fed lamb

SUMMARY:
This study will investigate the impact of consuming grass-finished lamb meat on blood omega-3 PUFAs and cardiovascular risk factors compared to concentrate-finished lamb meat. Healthy volunteers will consume three portions of lamb meat/week from a grass-finished meat treatment or a concentrate-finished meat treatment for four weeks. Blood samples will be taken at weeks zero and four. The primary outcome is to assess difference in change in omega-3 PUFA concentration in plasma and platelets between treatment groups. The secondary outcome is to assess between groups differences in change in cardiovascular disease risk factors including blood pressure, BMI and lipids among healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged between 18-64 years old.

Exclusion Criteria:

* Participants with a BMI of <18.5 km/m² and greater than >35 km/m².
* Participants who take prescribed medication, including statins to reduce LDL cholesterol, and any form of dietary supplements (excluding vitamin D).
* People who smoke.
* Participants who consume more than two portions of fish per month.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Fatty acid (%) change in blood plasma between treatments | Week 0 and week 4
  Primary outcome is to assess the impact of consuming grass vs concentrate finished lamb on blood plasma response in healthy volunteers
Fatty acid change (%) in blood plasma phospholipids between treatments | Week 0 and week 4
  Primary outcome is to assess the impact of consuming grass vs concentrate finished lamb on blood plasma phospholipid response in healthy volunteers

SECONDARY OUTCOMES:
Change in weight (kg) in participants between treatments | Week 0 and week 4
  Secondary outcome is to assess the impact of consuming grass vs concentrate finished lamb on weight among healthy volunteers
Change in Body Mass Index (BMI) in participants between treatments - calculated by dividing weight (kg) by height in meters squared | Week 0 and week 4
  Secondary outcome is to assess the impact of consuming grass vs concentrate finished lamb on weight and BMI response in healthy volunteers
Cholesterol | Week 0 and week 4
  Secondary outcome is to assess the impact of consuming grass vs concentrate finished lamb on total cholesterol, LDL, HDL and TAG response in healthy volunteers
Blood pressure (diastolic and systolic) | Week 0 and week 4
  Secondary outcome is to assess the impact of consuming grass vs concentrate finished lamb on blood pressure (diastolic and systolic) response in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Nigel D Scollan, PhD, Principal Investigator — Queen's University, Belfast; Jayne V Woodside, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- School of Biological Sciences, Queen's University Belfast, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perkins LS, Nugent AP, Woodside JV, Cardwell CR, Scollan ND. Consuming grass finished lamb improves blood plasma omega-3 fatty acid response among healthy consumers. Eur J Nutr. 2025 Jul 21;64(5):242. doi: 10.1007/s00394-025-03765-z. PMID 40690019

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT06607354/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT06607354/ICF_001.pdf